CLINICAL TRIAL: NCT06097403
Title: Prevalance of Cardiovascular Complications in Children With COVID 19 in Assuit University Children Hospital
Brief Title: Cardiovascular Complications in Children With COVID 19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Atif Abd Elhaleem, doctor, Assiut University
Other Study IDs: cardiovascular complications
Record Dates: First submitted 2023-10-22; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: COVID 19 Associated Coagulopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Covid 19 swap — diagnostic tool

SUMMARY:
Prevalance of cardiovascular complications in children with COVID 19 in Assuit university children hospital

DETAILED DESCRIPTION:
In December 2019, coronavirus disease 2019 (COVID-19) was first described in Wuhan, China, in patients complaining of flulike symptoms.1 The virus was isolated and identified as a new strain of coronavirus, now named SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2 ) . Cardiovascular complications of COVID-19 have received less medical attention; nevertheless, the first cases of myocarditis in COVID-19 patients have been reported,3, 4, 5, 6 and myocarditis has been recognized as the cause of death in some covid 19 patients.7 Pathology usually is focal within the myocardium, but there is a risk of arrhythmia as well as progression to fulminant heart failure and cardiogenic shock.

Clinical presentation of SARS-CoV-2 myocarditis varies among cases. Some patients may present with relatively mild symptoms, such as fatigue and dyspnea,4 , 5 whereas others report chest pain or chest tightness on exertion.3 , 6 Many patients do deteriorate, showing symptoms of tachycardia and acute-onset heart failure with cardiogenic shock.3, 4, 5 In these severe cases, patients may also present with signs of right-sided heart failure, including raised jugular venous pressure, peripheral edema, and right upper quadrant pain.10 The most emergent presentation is fulminant myocarditis, defined as ventricular dysfunction and heart failure within 2-3 weeks of contracting the virus.8 The early signs of fulminant myocarditis usually resemble those of sepsis: the patient often presents febrile with low pulse pressure, cold or mottled extremities, and sinus tachycardia.10 Myocarditis is an inflammatory disease of the heart characterized by inflammatory infiltrates and myocardial injury without an ischemic cause.8 The most commonly identifiable cause of myocarditis in the United States and other developed countries is viral.9 , Arrhythmia is recognized as one of the possible clinical manifestations of COVID-19 patients. One observational study of the clinical characteristics of COVID-19 patients in Hubei, China, reported a 7.3% incidence of heart palpitations among its 137 patients 13 Moreover, Wang et al reported that arrhythmia was a cause of intensive care unit transfer in 44.4% of COVID- Coagulation and inflammatory parameters are mildly altered in COVID-19 infection, whereas MIS-C is characterized by laboratory evidence of a proinflammatory and procoagulant state

ELIGIBILITY:
Inclusion Criteria:

* Patient less than 18 years old Presented with COVID 19

Exclusion Criteria:

* Not presented with covid19

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients with covid 19 confirmed with PCR from January 2023 till 31 december 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Prevalance of cardiovascular complications in children with COVID 19 | Baseline
  estimate the prevalence of cardiovascular complications among pediatric patients with covid 19 in Isolation Unit , Chest unit , and Cardiology unit in Assiut University Children Hospital

REFERENCES:
- [Background] Das BB, Akam-Venkata J, Abdulkarim M, Hussain T. Parametric Mapping Cardiac Magnetic Resonance Imaging for the Diagnosis of Myocarditis in Children in the Era of COVID-19 and MIS-C. Children (Basel). 2022 Jul 16;9(7):1061. doi: 10.3390/children9071061. PMID 35884045